CLINICAL TRIAL: NCT00774644
Title: The Objective of This Study is to Compare the Relative Bioavailability of Clarithromycin 500 mg Tablets (Ranbaxy Laboratories Limited) With That of BIAXIN® 500 mg Tablets in Healthy, Adult Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Clarithromycin 500mg Tablets Under Fasting Conditions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B025511
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): clarithromycin 500 mg tablets of Ranbaxy Laboratories Limited
  Interventions: Drug: Clarithromycin 500mg
- 2 (Active Comparator): BIAXIN® 500 mg tablets containing clarithromycin 500mg tablets
  Interventions: Drug: Clarithromycin 500mg

INTERVENTIONS:
Drug: Clarithromycin 500mg

SUMMARY:
The objective of this study is to compare the relative bioavailability of clarithromycin 500 mg tablets (Ranbaxy Laboratories Limited) with that of BIAXIN® 500 mg tablets in healthy, adult subjects under fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioavailability study on clarithromycin formulations comparing clarithromycin 500mg tablets of Ranbaxy Laboratories with Biaxin® tablets 500mg (containing clarithromycin 500 mg)in healthy, adult, human, male subjects under fasting conditions

Eligible subjects underwent pre-study examinations that included a physical examination, 12-lead ECG, and laboratory tests - including hematology, blood chemistries, urinalysis, infectious diseases (Hepatitis B, Hepatitis Ci HIV), and urine drugs of abuse. Laboratory testing for female subjects also included a serum pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Source of Subjects: Non-institutionalized subjects consisting of members of the community at large.
* Characterization of Study Group:

  1. All subjects selected for this study will be at least 18 years of age.
  2. Female subjects must be unable to become pregnant (postmenopausal for at least 1 year, or surgically sterile).
* Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process.
* At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.
* Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.
* Clinical laboratory measurements will include the following:

  * Hematology: hemoglobin, hematocrit,red blood cell count, platelets, and white blood cell count (with differential).

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma(during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested (including any penicillin product) should be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at check-in each study period. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drag within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant or who are able (women with child bearing potential).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-12; Primary Completion 2003-01 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Bioequiavlence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm